CLINICAL TRIAL: NCT03191162
Title: Phase II Clinical Trial for the Evaluation of Different Benznidazole Regimens for the Treatment of Chronic Chagas Disease in Adult Patients. Berenice Project
Brief Title: Evaluation of Different Benznidazole Regimens for the Treatment of Chronic Chagas Disease.
Acronym: MULTIBENZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-003789-21
Record Dates: First submitted 2017-06-08; First posted 2017-06-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Chagas Disease; Trypanosoma Cruzi Infection
Keywords: Benznidazole; PCR
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B300/60 (Active Comparator): Benznidazole 300mg/day p.o. divided in two doses for 60 days
  Interventions: Drug: Benznidazole
- B150/60 (Experimental): Benznidazole 150mg/day p.o. divided in two doses for 60 days
  Interventions: Drug: Benznidazole
- B400/15 (Experimental): Benznidazole 400mg/day p.o. divided in two doses for 15 days
  Interventions: Drug: Benznidazole

INTERVENTIONS:
Drug: Benznidazole — To evaluate different regimens of Benznidazole for the treatment of chronic Chagas disease
  Other Names: Abarax

SUMMARY:
A phase 2 clinical trial to evaluate the the efficacy of different benznidazole regimens (300mg/day for 60 days, 150mg/day for 60 days, and 400mg/day for 15 days) for the treatment of chronic Chagas disease in adult patients. The efficacy is assessed through the proportion of patients with negative parasitaemia measured by Polymerase Chain Reaction (PCR) during the first 12 months after starting treatment. The study will be performed in Spain, Brazil, Argentina and Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Diagnosis of Chagas disease through two different serological tests.
* Positive T. cruzi PCR in peripheral blood.
* Signed informed consent.

Exclusion Criteria:

* Previous treatment with Benznidazole or Nifurtimox.
* Alcohol consumption.
* Acute or chronic health problems that could interfere in the assessment of the efficacy or safety of the drug (acute infections, HIV infection, liver or renal impairment, etc).
* Nitroimidazole hipersensitivity.
* Concomitant or previous treatment with allopurinol or antifungal drugs.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with negative parasitaemia measured by PCR during the first 12 months after starting treatment | 12 months
  The treatment efficacy is assessed through the proportion of patients with negative parasitaemia measured by PCR during the first 12 months after starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Israel Molina, PhD, Principal Investigator — Hospital Universitario Vall d'Hebron Research Institute
Locations (7):
- Argentina (2):
  - Instituto Nacional de Parasitología Dr. Mario Fatala Chaben (ANLIS), Buenos Aires
  - Instituto de Cardiología de Corrientes Juana Francisca Cabral, Corrientes
- Brazil (2):
  - Centro de Pesquisas René Rachou - Fundação Oswaldo Cruz. (FIOCRUZ), Belo Horizonte
  - Hospital Universitário Clemente de Faria, Montes Claros
- Colombia (2):
  - Fundación Cardioinfantil - Instituto de Cardiología, Bogotá
  - Centro Atencion y Diagnóstico de Enfermedades Infecciosas, Bucaramanga
- Infectious Disease Department Vall d'Hebron Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bosch-Nicolau P, Fernandez ML, Sulleiro E, Villar JC, Perez-Molina JA, Correa-Oliveira R, Sosa-Estani S, Sanchez-Montalva A, Del Carmen Bangher M, Moreira OC, Salvador F, Mota Ferreira A, Eloi-Santos SM, Serre-Delcor N, Ramirez JC, Silgado A, Oliveira I, Martin O, Aznar ML, Ribeiro ALP, Almeida PEC, Chamorro-Tojeiro S, Espinosa-Pereiro J, de Paula AMB, Vaquiro-Herrera E, Tur C, Molina I; MULTIBENZ Study Group. Efficacy of three benznidazole dosing strategies for adults living with chronic Chagas disease (MULTIBENZ): an international, randomised, double-blind, phase 2b trial. Lancet Infect Dis. 2024 Apr;24(4):386-394. doi: 10.1016/S1473-3099(23)00629-1. Epub 2024 Jan 11. PMID 38218195
- [Derived] Molina-Morant D, Fernandez ML, Bosch-Nicolau P, Sulleiro E, Bangher M, Salvador F, Sanchez-Montalva A, Ribeiro ALP, de Paula AMB, Eloi S, Correa-Oliveira R, Villar JC, Sosa-Estani S, Molina I. Efficacy and safety assessment of different dosage of benznidazol for the treatment of Chagas disease in chronic phase in adults (MULTIBENZ study): study protocol for a multicenter randomized Phase II non-inferiority clinical trial. Trials. 2020 Apr 15;21(1):328. doi: 10.1186/s13063-020-4226-2. PMID 32293523